CLINICAL TRIAL: NCT02171416
Title: A Single-center, Double-blind Placebo-controlled Parallel Group Phase II Study of the Efficacy and Safety of Rilonacept in Subjects With Cold Contact Urticaria (CCU)
Brief Title: Cold Contact Urticaria Treatment With Rilonacept
Acronym: Cures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Karoline Krause, PD MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cures; 2012-005726-30 (EudraCT Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-24 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-03

CONDITIONS: Cold Contact Urticaria
MeSH Terms: conditions — Cold Urticaria | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo s.c every 7 days
  Interventions: Drug: Rilonacept
- Rilonacept 160mg (Experimental): Rilonacept s.c every 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilonacept
  Other Names: Arcalyst
  Arms: Placebo
Drug: Placebo
  Arms: Rilonacept 160mg

SUMMARY:
Cold contact urticaria (CCU) is a frequent form of physical urticaria that is characterized by the development of wheal and flare type skin reactions due to the release of histamine and other proinflammatory mast cell mediators following exposure of the skin to cold. Typically, symptoms occur within minutes after cold contact, including exposure to cold air, liquids or objects and are limited to cold exposed skin areas.

The investigators postulate that there is an overlap between acquired cold urticaria and cold-induced autoinflammatory syndromes, and that cold urticaria patients unresponsive to antihistamines will benefit from IL-1 targeting treatment strategies.

This study will evaluate the efficacy and safety of the IL-1 transfusion protein rilonacept in patients with cold contact urticaria who could not be successfully treated with first-line medication such as antihistamines.

This is a double-blind placebo-controlled parallel group phase II study of the efficacy and safety of rilonacept in subjects with CCU. A total of 20 patients will be included by the Urticaria specialty clinics of ACC. The total duration of the study course for each patient is 14 weeks and is divided in:

1. Screening period (2 weeks, days -14-0)
2. Placebo-controlled double-blind phase (Part A, 6 weeks, days 0-42)
3. Open label phase (Part B, 6 weeks, days 42-84) All eligible patients will be randomized (1:1 randomization) to one of two groups: 1) Rilonacept 160mg/week or 2) Placebo, and will receive the respective dose subcutaneously. Following the placebo-controlled double-blind phase patients will enter the open-label phase and receive rilonacept open-label treatment (160mg or 320mg depending on treatment response during part A).

ELIGIBILITY:
Inclusion Criteria:

* Adult ( > 18 years of age)
* Outpatients with CCU for more than six weeks. Urticaria symptoms must comprise wheal and itch and be resistant to conventional antihistamine treatment in standard doses
* Patients with a positive cold stimulation test at 4°C (assessed by TEMPtest 3.0)
* Informed consent signed and dated. Able to read, understand and willing to sign the informed consent form
* Able to read, understand and complete study-related questionnaires
* Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to self-administer SC injections or to have SC injections administered by a qualified person
* In women, negative pregnancy test
* Reliable method of contraception for both women of childbearing potential as well as men, during the course of the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* Subjects are considered eligible according to the following tuberculosis (TB) screening criteria:
* No history of latent or active TB prior to screening
* No signs or symptoms suggestive of active TB
* No recent close contacts with a person with active TB
* A negative QuantiFERON-TB test on day -14 (screening visit).

Exclusion Criteria:

* Treatment with a live (attenuated) virus vaccine during the month prior to day 0 (Randomization).
* A history of serious chronic or active infection(s) eg. listeriosis within six weeks prior to the screening visit.
* Evidence of acute or latent Tuberculosis as defined by the local guidelines/local medical practice
* A history of acute tuberculosis despite the proper treatment.
* Significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, metabolic, lymphatic or hematological disease that would adversely affect the subject's participation or evaluation in this study.
* Active systemic inflammatory condition including, but not limited to, rheumatoid arthritis, systemic lupus erythematosis, polymyalgia rheumatica, vasculitis, or myositis.
* History of fibromyalgia or chronic fatigue syndrome.
* Evidence of current HIV, Hepatitis B, or Hepatitis C infection by clinical or serological history.
* History of malignancies including malignant hematological disorders other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cervical cancer within five years of the Screening visit.
* Severe respiratory disease, including, but not limited to severe bronchiectasis, chronic obstructive pulmonary disease, bullous lung disease, uncontrolled asthma, or pulmonary fibrosis.
* Presence of any of the following laboratory abnormalities at enrollment visit: creatinine >1.5 x Upper Limit of Normal (ULN), WBC <3.6 x 103/mm3; platelet count <150,000 mm3; ALT or AST >2.0 x ULN.
* Previous ineffective treatment with IL1 inhibitor or other biologic agent.
* Known hypersensitivity to CHO cell derived therapeutics or proteins or any components of rilonacept.
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk.
* Present History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) that could limit the subject's ability to comply with study procedures.
* Lactating females or pregnant females.
* Enrollment in another investigational treatment or device study or use of an investigational agent, or no completion of less than 4 weeks or 5 half-lives, whichever is longer, since end of another investigational device or drug trial.
* Subjects for whom there is concern about compliance with the protocol procedures.
* Subjects who are detained officially or legally to an official institute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2018-02-28 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
To assess the effect of rilonacept on the clinical signs and symptoms of CCU | 6 weeks
  Change in symptom development (critical temperature thresholds (CTT) in CCU patients from baseline to day 42 in the rilonacept group as compared to the placebo group

SECONDARY OUTCOMES:
To assess the safety of rilonacept in subjects with CCU | 6 weeks
  This includes physical examination, routine safety laboratory assessments, vital signs and adverse event reporting

OTHER OUTCOMES:
Change in the patient's quality of life | 6 weeks
  Assessed by the Dermatology Life Quality Index (DLQI) from baseline to day 42 in the rilonacept group as compared to the placebo group and from baseline to the open-label treatment with rilonacept
Differences in mast cell mediator release | 6 weeks
  Measured in the blood of CCU patients during the challenge with cold water at day 42 in the rilonacept group as compared to the placebo group and during the open-label treatment in the rilonacept 160 mg group as compared to the 320 mg group

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Krause, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - University Berlin Charité ; Dermatology, Berlin
  - Universitätsmedizin, Mainz

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bonnekoh H, Butze M, Spittler S, Staubach P, Weller K, Scheffel J, Maurer M, Krause K. Inhibition of interleukin-1 with rilonacept is not effective in cold urticaria-Results of a randomized, placebo-controlled study. Clin Transl Allergy. 2023 Mar;13(3):e12226. doi: 10.1002/clt2.12226. PMID 36973954